CLINICAL TRIAL: NCT00695409
Title: A Phase II Study of Yttrium-90-Labeled Anti-CD20 Monoclonal Antibody in Combination With High-Dose Beam Followed by Autologous Stem Cell Transplantation for Poor Risk/Relapsed B-Cell Lymphoma
Brief Title: Yttrium-90 Ibritumomab Tiuxetan Plus High-Dose BEAM Followed By ASCT For Relapsed B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07076; P01CA030206 (NIH); P30CA033572 (NIH); CHNMC-07076; CDR0000597569 (Registry Identifier: NCI PDQ); NCI-2010-01231 (Registry Identifier: NCI CTPR)
Record Dates: First submitted 2008-06-10; First posted 2008-06-11 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Lymphoma
Keywords: recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Large-Cell, Immunoblastic | interventions — Rituximab; Carmustine; Cytarabine; Etoposide; Melphalan; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (RIT, ZBEAM, ASCT) (Experimental): RADIOIMMUNOTHERAPY: Patients receive yttrium Y 90 ibritumomab tiuxetan IV following rituximab IV on day -14. HIGH-DOSE COMBINATION CHEMOTHERAPY: Patients receive carmustine IV on days -7 and -6; etoposide IV over 1 hour twice daily and cytarabine IV over 2 hours twice daily on days -5 to -2; and melphalan IV on day -1. STEM CELL TRANSPLANTATION: Patients undergo autologous peripheral blood stem cell transplant on day 0. Patients also receive rituximab on day 8*. NOTE: * Some patients may also receive rituximab on day -1. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: carmustine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: ASCT; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: carmustine — Given IV
  Other Names: BCNU; BiCNU; bis-chloronitrosourea
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Procedure: ASCT — Undergo autologous peripheral blood stem cell transplant
  Other Names: Autologous Stem Cell Transplantation
Radiation: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan

SUMMARY:
This phase II clinical trial studies how well yttrium Y 90 ibritumomab tiuxetan, rituximab, and high-dose chemotherapy followed by peripheral blood stem cell transplant in treating patients with relapsed B-cell non-Hodgkin lymphoma. Monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan and rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Radiolabeled monoclonal antibodies can find tumor cells and carry tumor-killing substances to them without harming normal cells. Giving monoclonal antibody therapy, radioimmunotherapy (RIT), and high-dose combination chemotherapy before a peripheral blood stem cell transplant may be an effective treatment for non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the 2-year progression free survival.

SECONDARY OBJECTIVES:

II. To estimate the 2-year overall survival.

III. To estimate the 2-year cumulative incidence of progression.

IV. To estimate time to hematopoietic recovery, using absolute neutrophil and platelet engraftment.

V. To estimate incidence of grade 3-4 toxicities by Bearman Scale, Day 0 to Day 100.

VI. To estimate the response rate (CR/PR).

VII. To estimate 100-day treatment related mortality.

VIII. To estimate incidence of myelodysplasia and therapy related acute myeloid leukemia (AML).

IX. To descriptively compare the outcomes of patients treated on this protocol to a comparable patient population treated with chemotherapy alone.

OUTLINE: RADIOIMMUNOTHERAPY: Patients receive yttrium Y 90 ibritumomab tiuxetan intravenously (IV) following rituximab IV on day -14.

HIGH-DOSE COMBINATION CHEMOTHERAPY: Patients receive carmustine IV on days -7 and -6; etoposide IV over 1 hour twice daily (BID) and cytarabine IV over 2 hours BID on days -5 to -2; and melphalan IV on day -1.

STEM CELL TRANSPLANTATION: Patients undergo autologous peripheral blood stem cell transplant on day 0. Patients also receive rituximab on day 8*. NOTE: * Some patients may also receive rituximab on day -1. Treatment continues in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have biopsy proven diagnosis of low- and intermediate-grade non-Hodgkin lymphoma (NHL) working formulation B, C,D, E, F, and G; including mantle cell lymphoma; patients with transformed lymphoma are also eligible
* Demonstrated monoclonal CD20 positive b-cell population in lymph nodes and/or bone marrow
* Patients must have relapsed after achieving a complete or partial response to prior therapy, have never responded to prior therapy or have poor risk disease
* Patients with prior bone marrow involvement must have bone marrow aspiration and biopsy within 60 days prior to stem cell collection which shows =< 10% lymphomatous involvement of total cellularity; alternatively, patients with prior bone marrow involvement should have a normal bone marrow study which shows =< 10% lymphomatous involvement within 28 days before salvage chemotherapy
* Normal renal function test with serum creatinine of < upper limit of normal (ULN), and a creatinine clearance of >= 60 ml/min (measured or calculated)
* Adequate pulmonary function as measured by forced expiratory volume in 1 second (FEV1) > 60% of predicted measured, or a diffusion capacity of carbon monoxide (DLCO) >= 50% of predicted measured
* Cardiac ejection fraction of > 50% by echocardiogram or multi gated acquisition (MUGA) scan; the left ventricular ejection fraction (LVEF) from the prestudy echocardiogram (ECHO) or MUGA may be used for eligibility purposes, even if the prestudy stress test indicated a lower LVEF
* Adequate liver function tests with a bilirubin of =< 1.5 x ULN and serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) =< 2 x ULN
* Negative human immunodeficiency virus antibody
* Eastern Cooperative Oncology Group (ECOG) performance status = 0 or 1; karnofsky performance status (KPS) >= 80
* No active central nervous system (CNS) disease or prior history of CNS disease
* Patients must have recovered from last therapy and should be at least four weeks from prior radiation or systemic chemotherapy on the day of administration of Y2B8
* After the last systemic therapeutic chemotherapy (Cytoxan, administered only for stem cell mobilization is not considered therapeutic) and prior to initiation of high dose treatment, the patient should have a baseline computed tomography (CT) scan and positron emission tomography (PET) scan done; an fluorodeoxyglucose-computed tomography (FDG/CT) scan is sufficient, however, is clinically indicated, an additional diagnostic CT may be ordered; exception: if scans were done and were negative for disease just prior to priming chemotherapy (therapeutic or nontherapeutic) and subsequent stem cell harvest, they do not need to be repeated prior to initiation of high dose treatment

Exclusion Criteria:

* Presence of human anti-Zevalin antibody (HAZA)
* Prior radioimmunotherapy
* Failure to collect adequate number of CD34+ cells >= 3 x 10^6/kg
* Abnormal cytogenetic study not related to the underlying lymphoma on the bone marrow aspirate sample prior to stem cell collection; if cytogenetics were not performed on the marrow aspirate prior to stem cell collection, cytogenetics on the peripheral blood may be performed
* Prior bone marrow transplantation
* Prior malignancy except for:

  * Adequately treated basal cell or squamous cell skin cancer
  * Adequately treated noninvasive carcinoma
  * Other cancer from which the patient has been disease-free for at least five years
* Active evidence of Hepatitis B or C infection; Hepatitis B surface antigen positive
* Patients who have had prior radiation to the lung will be excluded from the study, although mediastinal irradiation will be permitted if minimal lung is in the treatment volume
* Patients who have received > 500cGy radiation to the kidneys will be excluded from the study
* Patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-03-18 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Y. Krishnan, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Started | 122
Completed | 122
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 104
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 122

OUTCOME MEASURES:

1. Primary Outcome: 2-Year Progression-Free Survival
Description: Progression-free survival (PFS) was defined as time from peripheral stem cell infusion to recurrence, progression or death. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works. Progression-free survival was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula [Breslow NE, Day NE. Statistical methods in cancer research: volume II, the design and analysis of cohort studies. IARC Sci Publ 1987;82:1-406.]
Time Frame: From peripheral stem cell infusion (Day0 ASCT) to first observation of progressive disease or death due to any cause, whichever comes first, assessed up to 5 years
Population: 6 patients did not receive full treatment so are excluded from the result analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 116
Percentage of Participants (%) | 71 [61 to 78]

2. Secondary Outcome: 2-Year Overall Survival
Description: Overall survival (OS) was measured from peripheral stem cell infusion to death from any cause. It was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula. [Breslow NE, Day NE. Statistical methods in cancer research: volume II, the design and analysis of cohort studies. IARC Sci Publ 1987;82:1-406.]
Time Frame: From peripheral stem cell infusion (Day0 ASCT) to death due to any cause, assessed up to 5 years
Population: 6 patients did not receive full treatment so are excluded from the result analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 116
Percentage of Participants (%) | 89 [82 to 94]

3. Secondary Outcome: 2-Year Cumulative Incidence of Progression
Description: The cumulative incidence was estimated after taking into account the competing risk of early death.
Time Frame: From peripheral stem cell infusion (Day0 ASCT) to date of first observation of progressive disease or relapsed disease, assessed up to 5 years
Population: 6 patients did not receive full treatment so are excluded from the result analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 116
Percentage of Participants (%) | 28 [20 to 37]

4. Secondary Outcome: Number of Patients With Active Disease at ASCT Achieving CR/PR by Day 100 After ASCT
Description: Responses are assessed using the Revised Criteria for Malignant Lymphoma Response Definitions for Clinical Trials (Cheson et al. 2007). Complete Response (CR) defined as disappearance of all evidence of disease. Partial Response (PR) defined as regression of measurable disease and no new sites.
Time Frame: Up to Day 100 post-ASCT
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Active Disease at ASCT: Patients receiving the full treatment (RIT/ZBEAM) with active disease at time of ASCT
Arm/Group | Patients With Active Disease at ASCT
Number analyzed (Participants) | 64
Participants | 53

5. Secondary Outcome: Number of Patients With Grade 3-4 Bearman Toxicities.
Description: Toxicities were recorded using the modified Bearman Scale for non-hematologic adverse events.
Time Frame: From initial of study treatment to Day 100 post-ASCT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 122
Participants
  Gastrointestinal Toxicity | 1
  Pulmonary Toxicity | 1
  No Grade 3-4 Toxicity | 120

6. Secondary Outcome: 100-Day Treatment-Related Mortality
Description: The cumulative incidence was estimated after taking into account the competing risk of relapse post-ASCT.
Time Frame: From peripheral stem cell infusion (Day0 ASCT) to death due to any couse, assessed up to 5 years
Population: 6 patients did not receive full treatment so are excluded from the result analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants (%)
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 116
Percentage of Participants (%) | 0.9 [0.1 to 6.1]

7. Secondary Outcome: Time to Neutrophil Recovery
Description: Neutrophil recovery was defined as the first of 3 consecutive days of an absolute neutrophil count ≥ 500/µL.
Time Frame: From peripheral stem cell infusion (Day0 ASCT) till the first of 3 consecutive days of an absolute neutrophil count ≥ 500/µL.)
Population: 6 patients did not receive full treatment so are excluded from the result analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 116
Days | 10 [9 to 13]

8. Secondary Outcome: Time to Platelet Recovery
Description: Platelet recovery was defined as the first of 7 consecutive days with a platelet count ≥ 20,000/µL with no transfusions.
Time Frame: From peripheral stem cell infusion (Day0 ASCT) till the first of 7 consecutive days with a platelet count ≥ 20,000/µL with no transfusions
Population: 6 patients did not receive full treatment so are excluded from the result analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 116
Days | 12 [8 to 86]

9. Secondary Outcome: Number of Patients With RIT/ZBEAM Developing Therapy Induced MDS and AML
Description: Patient receiving the full treatment of RIT/ZBEAM developed therapy induced MDS or AML.
Time Frame: From peripheral stem cell infusion (Day0 ASCT) to onset of therapy induced MDS/AML, assessed up to 5 years
Population: 6 patients did not receive full treatment so are excluded from the result analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
Number analyzed (Participants) | 116
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Treatment (RIT, ZBEAM, ASCT)
All-Cause Mortality (participants affected / at risk) | 25/122
Serious Adverse Events (participants affected / at risk) | 2/122
Other Adverse Events (participants affected / at risk) | 121/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (RIT, ZBEAM, ASCT) (N=122)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Secondary Malignancy (Nervous system disorders) | 1 (1) — Neuroendocrine Cancer
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (RIT, ZBEAM, ASCT) (N=122)
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 2/121 (2)
Bone marrow cellularity (Blood and lymphatic system disorders) | 11/121 (11)
Hemoglobin (Blood and lymphatic system disorders) | 119/121 (119)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 117/121 (130)
Lymphopenia (Blood and lymphatic system disorders) | 118/121 (129)
Myelodysplasia (Blood and lymphatic system disorders) | 1/121 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 115/121 (154)
Phlebitis (including superficial thrombosis) (Blood and lymphatic system disorders) | 1/121 (1)
Platelets (Blood and lymphatic system disorders) | 115/121 (121)
Thrombosis/embolism (vascular access-related) (Blood and lymphatic system disorders) | 1/121 (1)
Thrombosis/thrombus/embolism (Blood and lymphatic system disorders) | 2/121 (4)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 2/121 (2)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 4/121 (4)
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 3/121 (3)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 13/121 (17)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 2/121 (2)
Hypertension (Cardiac disorders) | 36/121 (43)
Hypotension (Cardiac disorders) | 47/121 (47)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1/121 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 18/121 (18)
Palpitations (Cardiac disorders) | 3/121 (3)
Pericardial effusion (non-malignant) (Cardiac disorders) | 5/121 (5)
Prolonged QTc interval (Cardiac disorders) | 19/121 (19)
Pulmonary hypertension (Cardiac disorders) | 1/121 (1)
Right ventricular dysfunction (cor pulmonale) (Cardiac disorders) | 1/121 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 44/121 (56)
Valvular heart disease (Cardiac disorders) | 4/121 (4)
Ventricular arrhythmia (Cardiac disorders) | 2/121 (2)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 4/121 (4)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 7/121 (10)
Tinnitus (Ear and labyrinth disorders) | 8/121 (8)
Endocrine - Other (Specify, __) (Endocrine disorders) | 1/121 (1)
Hot flashes/flushes (Endocrine disorders) | 2/121 (2)
Dry eye syndrome (Eye disorders) | 5/121 (5)
Glaucoma (Eye disorders) | 2/121 (2)
Nystagmus (Eye disorders) | 3/121 (3)
Ocular surface disease (Eye disorders) | 3/121 (3)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 6/121 (8)
Retinal detachment (Eye disorders) | 1/121 (1)
Vision-blurred vision (Eye disorders) | 7/121 (7)
Vision-flashing lights/floaters (Eye disorders) | 2/121 (2)
Watery eye (epiphora, tearing) (Eye disorders) | 3/121 (3)
Anorexia (Gastrointestinal disorders) | 100/121 (100)
Colitis (Gastrointestinal disorders) | 8/121 (8)
Constipation (Gastrointestinal disorders) | 68/121 (69)
Dehydration (Gastrointestinal disorders) | 8/121 (8)
Diarrhea (Gastrointestinal disorders) | 111/121 (112)
Distension/bloating, abdominal (Gastrointestinal disorders) | 31/121 (31)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 48/121 (48)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 16/121 (16)
Esophagitis (Gastrointestinal disorders) | 7/121 (7)
Fistula, GI (Gastrointestinal disorders) | 1/121 (1)
Flatulence (Gastrointestinal disorders) | 6/121 (6)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1/121 (1)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 8/121 (9)
Heartburn/dyspepsia (Gastrointestinal disorders) | 37/121 (37)
Hemorrhoids (Gastrointestinal disorders) | 18/121 (18)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 2/121 (2)
Incontinence, anal (Gastrointestinal disorders) | 1/121 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 101/121 (152)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 98/121 (151)
Nausea (Gastrointestinal disorders) | 113/121 (114)
Obstruction, GI (Gastrointestinal disorders) | 1/121 (1)
Proctitis (Gastrointestinal disorders) | 1/121 (1)
Salivary gland changes/saliva (Gastrointestinal disorders) | 11/121 (11)
Stricture/stenosis (including anastomotic), GI (Gastrointestinal disorders) | 1/121 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 37/121 (37)
Vomiting (Gastrointestinal disorders) | 94/121 (96)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 118/121 (120)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 32/121 (32)
Insomnia (General disorders) | 72/121 (72)
Pain (General disorders) | 116/121 (646)
Pain - Other (Specify, __) (General disorders) | 34/121 (42)
Rigors/chills (General disorders) | 49/121 (49)
Sweating (diaphoresis) (General disorders) | 20/121 (20)
Weight gain (General disorders) | 34/121 (34)
Weight loss (General disorders) | 61/121 (61)
Hematoma (Blood and lymphatic system disorders) | 3/121 (3)
Hemorrhage, GI (Blood and lymphatic system disorders) | 33/121 (35)
Hemorrhage, GU (Blood and lymphatic system disorders) | 24/121 (26)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 23/121 (24)
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 2/121 (2)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 36/121 (36)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4/121 (4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 6/121 (6)
Allergy/Immunology - Other (Specify, __) (Immune system disorders) | 1/121 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 8/121 (8)
Febrile neutropenia (Infections and infestations) | 39/121 (40) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 28/121 (32) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 47/121 (60)
Infection with unknown ANC (Infections and infestations) | 13/121 (15)
Edema:head and neck (General disorders) | 13/121 (13)
Edema:limb (General disorders) | 52/121 (52)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 60/121 (60)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 71/121 (71)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 2/121 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 106/121 (106)
Alkaline phosphatase (Metabolism and nutrition disorders) | 41/121 (41)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1/121 (1)
Amylase (Metabolism and nutrition disorders) | 1/121 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 23/121 (23)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 12/121 (13)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 5/121 (5)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 92/121 (92)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 43/121 (43)
Creatinine (Metabolism and nutrition disorders) | 14/121 (14)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 70/121 (78)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 48/121 (48)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 8/121 (8)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 36/121 (36)
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 1/121 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 47/121 (49)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5/121 (5)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 82/121 (84)
Proteinuria (Metabolism and nutrition disorders) | 2/121 (2)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 5/121 (5)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 103/121 (103)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 34/121 (34)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 7/121 (8)
Obesity (Metabolism and nutrition disorders) | 76/121 (190)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 3/121 (3)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 2/121 (2)
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 2/121 (2)
Joint-effusion (Musculoskeletal and connective tissue disorders) | 1/121 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 1/121 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 84/121 (123)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 3/121 (3)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1/121 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2/121 (2)
Arachnoiditis/meningismus/radiculitis (Nervous system disorders) | 1/121 (1)
Ataxia (incoordination) (Nervous system disorders) | 2/121 (2)
Cognitive disturbance (Nervous system disorders) | 1/121 (1)
Confusion (Nervous system disorders) | 18/121 (18)
Dizziness (Nervous system disorders) | 66/121 (66)
Encephalopathy (Nervous system disorders) | 2/121 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 17/121 (17)
Memory impairment (Nervous system disorders) | 7/121 (7)
Mood alteration (Nervous system disorders) | 88/121 (137)
Neurology - Other (Specify, __) (Nervous system disorders) | 10/121 (10)
Neuropathy: cranial (Nervous system disorders) | 1/121 (1)
Neuropathy: motor (Nervous system disorders) | 7/121 (8)
Neuropathy: sensory (Nervous system disorders) | 42/121 (43)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 12/121 (12)
Seizure (Nervous system disorders) | 2/121 (2)
Somnolence/depressed level of consciousness (Nervous system disorders) | 7/121 (8)
Syncope (fainting) (Nervous system disorders) | 3/121 (4)
Tremor (Nervous system disorders) | 6/121 (6)
Cystitis (Renal and urinary disorders) | 1/121 (1)
Incontinence, urinary (Renal and urinary disorders) | 3/121 (3)
Renal failure (Renal and urinary disorders) | 2/121 (2)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 3/121 (3)
Stricture/stenosis (including anastomotic), GU (Renal and urinary disorders) | 1/121 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 11/121 (11)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1/121 (1)
Urine color change (Renal and urinary disorders) | 8/121 (8)
Erectile dysfunction (Reproductive system and breast disorders) | 3/121 (3)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 2/121 (2)
Libido (Reproductive system and breast disorders) | 2/121 (2)
Sexual/Reproductive Function - Other (Specify, __) (Reproductive system and breast disorders) | 1/121 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1/121 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 17/121 (17)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 9/121 (9)
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 59/121 (61)
Cough (Respiratory, thoracic and mediastinal disorders) | 72/121 (73)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 35/121 (35)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 25/121 (25)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 9/121 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 20/121 (20)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1/121 (1)
Obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 1/121 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 11/121 (11)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 21/121 (23)
Pulmonary fibrosis (radiographic changes) (Respiratory, thoracic and mediastinal disorders) | 1/121 (1)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 54/121 (74)
Vital capacity (Respiratory, thoracic and mediastinal disorders) | 27/121 (27)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 11/121 (11)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Investigations) | 6/121 (6)
Syndromes - Other (Specify, __) (Investigations) | 9/121 (9)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 14/121 (14)
Burn (Skin and subcutaneous tissue disorders) | 1/121 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 24/121 (27)
Dry skin (Skin and subcutaneous tissue disorders) | 29/121 (30)
Flushing (Skin and subcutaneous tissue disorders) | 35/121 (35)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 50/121 (50)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 21/121 (21)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 1/121 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1/121 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1/121 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 46/121 (46)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 84/121 (84)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 8/121 (8)
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 3/121 (3)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1/121 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1/121 (1)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 6/121 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT00695409/Prot_SAP_000.pdf